CLINICAL TRIAL: NCT07145268
Title: Clinical Study to Evaluate the Possible Antifibrotic Effect of Zinc Sulphate in Chronic HBV Patient Receiving Anti Viral Therapy
Brief Title: Zinc Sulphate in Treatment Fibrosis in HBV Patient Receiving Antiviral Therapy
Acronym: HBV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Ahmed Mohamed Ragai Elrefaey, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zinc sulphate in HBV
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Liver Fibroses; HBV (Hepatitis B Virus)
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B | interventions — entecavir; Zinc; Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (control group) (Placebo Comparator): 22 patients will continue their standard antiviral therapy (Entecavir 0.5 mg) for 6 months.
  Interventions: Drug: Entecavir (ETV)
- (zinc group) (Active Comparator): 22 patients will receive Zinc suIphate 220 mg orally once daily (equivalent to 50 mg elemental zinc), in addition to their standard antiviral therapy (Entecavir 0.5 mg), for 6 months.
  Interventions: Drug: Zinc (zinc sulphate)

INTERVENTIONS:
Drug: Entecavir (ETV) — Standard antiviral therapy with Entecavir 0.5 mg orally once daily for 6 months."(control group)
  Arms: (control group)
Drug: Zinc (zinc sulphate) — Zinc sulfate 220 mg orally once daily (50 mg elemental zinc) in addition to Entecavir 0.5 mg, for 6 months."
  Arms: (zinc group)

SUMMARY:
This study aims to investigate the possible safety and efficacy of Zinc sulphate as antifibrotic agent in chronic HBV patient receiving antiviral therapy.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a serious public health problem worldwide and major cause of chronic hepatitis, fibrosis, cirrhosis, and hepatocellular carcinoma (HCC). It was estimated that approximately 2 billion people have serological evidence of past or present HBV infection. More than 350 million are chronic carriers of HBV. (1)

Chronic hepatitis B describes a spectrum of disease usually characterized by the presence of detectable hepatitis B surface antigen (HBsAg) in the blood or serum for longer than 6 months. In some people, chronic hepatitis B is inactive and does not present significant health problems, but others may progress to liver fibrosis, cirrhosis and HCC. (1)

Liver fibrosis due to viral or metabolic chronic liver diseases is a major challenge of global health. Correlating with liver disease progression, fibrosis is a key factor for liver disease outcome and risk of HCC. (2)

Removal or elimination of the causative agent such as control or cure of viral infection has shown that liver fibrosis is reversible. There is a huge unmet medical need for anti-fibrotic therapies to prevent liver disease progression and HCC development. (2) Liver fibrosis is the excessive accumulation of extracellular matrix proteins including collagen that occurs in most types of chronic liver diseases. In the case of chronic HBV infection, ongoing liver inflammation and immune-mediated damage led to fibrosis over time. (2) Zinc is an essential trace element required for normal cell growth, development, and differentiation. It is involved in DNA synthesis, RNA transcription, and cell division and activation. It is a critical component in many zinc protein/enzymes, including critical zinc transcription factors. Zinc deficiency/altered metabolism is observed in many types of liver disease, including alcoholic liver disease and viral liver disease. (3) Serum zinc levels are significantly decreased in patients with acute hepatitis B infection and are frequently depressed with HBV cirrhosis (similar to HCV cirrhosis). Specifically designed zinc finger proteins had been used in an attempt to inhibit HBV viral transcription with some success, and this is a potential therapeutic target for new HBV drugs. Importantly, marginal zinc deficiency appears to impair the efficacy of hepatitis B vaccination. This is another example of how zinc deficiency may impair immune function with special relevance to liver disease. (3) Zinc supplementation suppresses the progression of liver fibrosis induced by bile duct ligation in mice. (4) Liver biopsy is recognized as the gold standard for disease monitoring; however, the procedure is invasive and bedeviled with potential complications. For these reasons, non-invasive biomarkers of fibrosis are now being evaluated as alternatives to liver biopsy. (5) Fibronectin is a glycoprotein involved in wound healing and extracellular matrix formation. Elevated levels are associated with liver fibrosis due to increased extracellular matrix deposition. It reflects fibrogenesis activity and can serve as an early indicator of fibrotic progression or regression. (6) Serum hyaluronic acid (HA) level is a precise predictor of extensive liver fibrosis in chronic hepatitis B. Stage of fibrosis is well correlated with HA which can reflect the severity of fibrosis. Thus, it can be used as a noninvasive test to monitor these patients. (7)

ELIGIBILITY:
Inclusion Criteria:

* Patients with fibrosis stage (F2&F3) post chronic HBV infection receiving standard antiviral therapy.
* Age > 18 and < 65 years.

Exclusion Criteria:

* Patients with prior history of liver transplantation.
* Patients with prior history of hepatocellular carcinoma.
* Patients coinfected with HIV or HCV.
* Patients with any malignancies.
* Pregnant and lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in fibrosis scores. | 6 months

SECONDARY OUTCOMES:
Change in serum biomarkers | 6 months
  The secondary outcome is decrease in serum levels of the measured biological markers which are (fibronectin & HA)